CLINICAL TRIAL: NCT04523688
Title: Vaccination With Autologous Dendritic Cells Loaded With Autologous Tumour Homogenate in Glioblastoma: a Phase II Study
Brief Title: Vaccination With Autologous Dendritic Cells Loaded With Autologous Tumour Homogenate in Glioblastoma
Acronym: Combi G-Vax
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST191.05
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2024-09

CONDITIONS: Glioblastoma; Vaccination
Keywords: glioblastoma; dendritic cells; vaccine; temozolomide; Stupp regimen; cellular therapy
MeSH Terms: conditions — Glioblastoma | interventions — Vaccines; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental treatment (Experimental): Induction phase: 4 weekly doses of dendritic cell vaccine (10x10exp6 cells) intradermally administered (weeks 1-4).
  Maintenance phase: 28 days cycles with vaccine administration (start on week 7) and adjuvant temozolomide (150-200mg/m2/day) assumed orally from day 1 to 5 q28 (start on week 5). The combined maintenance treatment will continue until disease progression, unacceptable toxicity or withdrawal of consent by the patient, or up to a maximum of 1 year of treatments.
  After disease progression or the end of maintenance phase, is foreseen a one-year follow-up phase for each subject.
  Interventions: Biological: Autologous Dendritic Cells (DC) vaccine; Drug: Temozolomide

INTERVENTIONS:
Biological: Autologous Dendritic Cells (DC) vaccine — 10×10exp6 autologous dendritic cells loaded with autologous tumour homogenate given by intradermal injection (day 1)
Drug: Temozolomide — Adjuvant temozolomide assumed orally from day 1 to 5 (start on week 5). Dosage: 150mg/m2/day for the first cycle and 200 mg/m2/day for subsequent cycles (q28).

SUMMARY:
Single arm, monocentric trial to assess the safety and the progression-free survival related to the combined treatment of dendritic cell vaccine loaded with autologous tumor homogenate and temozolomide in patients operated for glioblastoma and then treated with standard radiochemotherapy (according to Stupp regimen).

DETAILED DESCRIPTION:
Single arm, monocentric trial to assess the safety and the progression-free survival related to the combined treatment of dendritic cell vaccine loaded with autologous tumor homogenate and temozolomide in patients operated for glioblastoma and then treated with standard radiochemotherapy (according to Stupp regimen).

The experimental treatment consists of an induction phase with 4 weekly doses of dendritic cell vaccine (10x10exp6 cells) intradermally administered (weeks 1-4), followed by a maintenance phase consisting of 28 days cycles with vaccine administration (start on week 7) and adjuvant temozolomide (150-200mg/m2/day) assumed orally from day 1 to 5 q28 (start on week 5). The combined maintenance treatment will continue until disease progression, unacceptable toxicity or withdrawal of consent by the patient, or up to a maximum of 1 year of treatments. After disease progression or the end of maintenance phase, is foreseen a one-year follow-up phase for each subject.

Primary objectives are clinical activity and safety of the study treatment. Secondary objectives are the evaluation of the prognostic role of the positive Delayed-Type Hypersensitivity (DTH) skin test after at least four vaccine administrations, the OS and the immunological efficacy of the study treatment. A series of exploratory objectives will be also assessed on samples from patients who participate to this optional part of the trial.

Simon's two-stage design (Simon, 1989) will be used for the sample size calculation.

A planned interim analysis will be done after the recruitment of the first 9 evaluable patients for toxicity and for efficacy.

If study will not be stopped due to lack of safety or efficacy, a total of 28 evaluable patients will be enrolled for the trial.

Time to events (PFS and OS) will be calculated with the Kaplan-Meier method and the analysis was performed on the eligible population. For the primary objective, the proportion of patients without progression at three months from leukapheresis date will be evaluated. The proportion of patients experiencing vaccine-related grade ≥ 3 adverse events (AEs) during the treatment will be inferred by means of the two-sided Clopper-Pearson, or a more appropriate one, 95% confidence interval. Descriptive statistics will be used to assess the extent of the secondary endpoints.

ELIGIBILITY:
After signing the informed consent form for pre-screening, patient will assess the procedures to obtain sufficient leukapheretic material for the dendritic cell vaccine manufacturing and will perform the standard radiochemotherapy treatment (Stupp regimen) for the disease.

For the pre-screening phase of the study the eligibility criteria are:

1. Histologically confirmed "monofocal" glioblastoma
2. Near-complete resection (= 5 ml residual tumor volume) confirmed by "central neuroradiologist on magnetic resonance imaging (MRI) or CT scan within 72 h postoperative"
3. Karnofsky performance status (KPS) = 70% or performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale (Appendix A)
4. Be willing and able to provide written informed consent/assent for the pre-screening phase of the trial.
5. Be = 18 years of age on day of signing informed consent.
6. Life expectancy of greater than 12 weeks.
7. Patient suitable for the collection of biological material from leukapheresis:

   serological tests HIV, hepatitis B virus (HBV), HCV, Treponema pallidum negative; normal cardiological parameters (ECG and cardiological examination); evaluation by transfusionist to exclude possible contraindications to leukapheresis.
8. Patient candidate to standard radiochemotherapy (Stupp regimen)
9. Appropriate 12-lead ECG and echocardiogram.

After pre-screening, patient will be enrolled based on subsequent Inclusion Criteria:

1. Histologically confirmed "monofocal" glioblastoma
2. THE AUTOLOGOUS SURGICAL SPECIMEN NEEDED FOR VACCINE MANUFACTURING MUST HAVE BEEN COLLECTED AND SENT TO THE SOMATIC CELL THERAPY LAB OF ISTITUTO SCIENTIFICO ROMAGNOLO PER LO STUDIO E LA CURA DEI TUMORI (IRST) ISTITUTO DI RICOVERO E CURA A CARATTERE SCIENTIFICO (IRCCS) AND MUST FULFIL ALL THE ACCEPTANCE CRITERIA PRESCRIBED BY THE GOOD MANUFACTURING PRACTICES (GMP) PROCEDURES.
3. Availability of sufficient leukapheretic material for the preparation of the vaccine product.
4. No progressive disease near-complete resection (= 5 ml residual tumor volume) confirmed by MRI after standard radiochemotherapy treatment (Stupp regimen)
5. Patients must have recovered (grade 1 or less by CTCAE 5.0) from all the events related to previous treatments.
6. Be willing and able to provide written informed consent/assent for the trial.
7. Be >= 18 years of age on day of signing informed consent.
8. Have a Karnofsky performance status (KPS) = 70% or a performance status of 0 or 1 on the ECOG Performance Scale.
9. Demonstrate adequate organ and marrow function

Exclusion Criteria:

1. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy > 10 mg prednisone equivalent or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
2. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
3. Has a known history of active Bacillus Tuberculosis (TB)
4. Previous treatment with a cancer vaccine
5. Other known malignant neoplastic diseases in the patient's medical history with a disease-free interval of less than 5 years, except basal or squamous cell carcinoma of the skin and in situ carcinoma of the cervix uteri treated with radical surgery.
6. Any known history of or is positivity of any serologic marker indicative of infection by Treponema pallidum, hepatitis B virus (HBsAg, HBsAb, HBcAB), hepatitis C virus (HCVAb, HCV RNA quantitative), human immunodeficiency virus (HIV), whether actual or previous.
7. Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
clinical activity | about 55 months
  Progression free survival (PFS), measured as the proportion of patients without progression of disease at three months from leukapheresis
Incidence of Treatment-Emergent Adverse Events | about 55 months
  Proportion of patients experienced grade 3 or higher adverse events related to the study treatment

SECONDARY OUTCOMES:
Immune response in vivo | about 32 months
  Evaluation of the prognostic role of a positive DTH test after at least four vaccine administrations
Clinical Outcome (Overall Survival (OS)) | about 55 months
  Overall Survival (OS) is calculated as the time from the date of leukapheresis to the date of death for any cause. Patients still alive at the time of analysis are censored at the last time they are known to be alive.
Immunological efficacy | about 55 months
  Immunological efficacy: ability to enhance the proportion of circulating immune effectors specific for tumor antigens; evaluation of the persistence of an anti-tumor immune response; determination of plasma levels of a panel of inflammatory cytokines and pro-angiogenic factors; evaluation of the prognostic and predictive role of tumor antigen expression in tumor tissue; analysis of the prognostic and predictive role of immune cells in the peripheral blood and in the tumor microenvironment
Human leukocyte antigen (HLA) class I and II characterization characterization of patients | about 32 months
  Explorative endpoint (optional participation for patients): HLA class I and II characterization of patients

CONTACTS AND LOCATIONS:
Overall Officials: Laura Ridolfi, DR, Study Chair — IRST IRCCS
Locations (1):
- Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, FC, Italy